CLINICAL TRIAL: NCT03886090
Title: Facilitating Motor Skill Learning by Aerobic Training in Parkinson's Disease II
Brief Title: Facilitating Motor Skill Learning in Parkinson's Disease II (FaST-PD II)
Acronym: FaST-PD II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg (Other)
Collaborators: German Foundation for Neurology (Other); Department of Molecular Neurology, Faculty of Medicine, University Erlangen-Nürnberg (Other); Klinik für Neurologie, Krankenhaus Rummelsberg (Unknown)
Responsible Party: Principal Investigator, Simon Steib, PhD, Principal Investigator, University of Erlangen-Nürnberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DSN-2018
Record Dates: First submitted 2019-03-20; First posted 2019-03-22 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; motor learning; neuroplasticity; aerobic exercise; cardiovascular exercise; balance; postural instability; motor memory; consolidation
MeSH Terms: conditions — Parkinson Disease | interventions — Exercise; RE1-silencing transcription factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- motor skill practice + aerobic exercise (Experimental): acute bout of aerobic exercise following motor skill practice
  Interventions: Behavioral: aerobic exercise; Behavioral: motor learning
- motor skill practice + rest (Active Comparator): seated rest following motor skill practice
  Interventions: Behavioral: rest; Behavioral: motor learning

INTERVENTIONS:
Behavioral: aerobic exercise — Single-bout of moderate intensity aerobic exercise on a cycle ergometer following motor skill practice
  Arms: motor skill practice + aerobic exercise
Behavioral: rest — Seated rest following motor skill practice
  Arms: motor skill practice + rest
Behavioral: motor learning — Motor learning task on a stability platform (Stabilometer). Participants try to keep the tiltable platform in a horizontal position.

SUMMARY:
The study is designed to assess the effects of cardiovascular (aerobic) exercise on motor skill learning in Parkinson patients. Specifically, the investigators examine whether a single bout of moderate-intense aerobic exercise, performed immediately following motor skill practice, facilitates motor memory consolidation. In this experimental trial, participants will be randomly allocated to either an intervention group (motor skill practice + aerobic exercise) or control group (motor skill practice + seated rest).

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a progressive neurodegenerative disorder that is characterized by motor control impairments, such as gait disturbances and postural instability. Beneficial effects of exercise are attributed to mechanisms of neuroplasticity, and task-specific motor training (repeated practice of a skill) is consequently considered to be a motor learning process. Importantly, the formation (acquisition) and consolidation of motor memories is impaired in PD compared to healthy individuals of similar age.

Thus, it is crucial to identify strategies to enhance motor learning in people with PD. Recent studies have accumulated evidence to show that acute (single bouts of) cardiovascular exercise can facilitate motor skill learning. However, this evidence is mainly derived from studying healthy individuals. In a first study including PD patients, we recently found improved motor memory consolidation, but not skill acquisition, when practice was preceded by a single bout of cardiovascular exercise.

These results suggest that acute exercise may enhance motor memory formation processes, but could potentially interfere with motor skill acquisition when performed prior to practice. Consequently, the present study investigates whether performing a single bout of cardiovascular exercise immediately following skill practice will enhance motor memory consolidation without affecting skill acquisition in PD.

In an experimental trial, participants will be randomly allocated to one of two groups. Both groups will practice balancing on a stability platform (motor learning task). The experimental group will additionally perform a bout of aerobic exercise (cycle ergometer) immediately following motor practice, while the control group will rest. Subsequently, motor skill retention will be tested after 24 hour and seven-days.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease stage 1-3 on Hoehn & Yahr scale
* Ability to stand unaided and walk without an assistive device
* Stable medication during the study period
* Unfamiliar to the motor learning task

Exclusion Criteria:

* On-off and wearing-off phenomena
* Unstable medical or psychiatric illness
* Clinically relevant cardiovascular or orthopaedic disease
* Severe polyneuropathy
* Cognitive impairment
* Smoking > 10 cigarettes/day
* Caffeine > 6 cups of coffee/day
* Alcohol > 50 g (two glasses)/day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2020-02-24 (Actual)

PRIMARY OUTCOMES:
Time in balance | Day 1: performance at end of skill acquisition (last practice block), Day 2: 24-hour retention performance, Day 3: seven-day retention performance
  Motor memory consolidation: Change of time in balance (angular displacement ±5° from horizontal) from skill practice (last block of skill acquisition) to 24-hour and seven-day retention test.

SECONDARY OUTCOMES:
Root mean square error (RMSE) | Day 1: performance at end of skill acquisition (last practice block), Day 2: 24-hour retention performance, Day 3: seven-day retention performance
  Memory consolidation: Change of root mean square error (average angular deviation from horizontal) from skill practice (last block of skill acquisition) to one-day and seven-day retention test.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Steib, Dr., Principal Investigator — Friedrich-Alexander University Erlangen-Nürnberg, Department of Sport Science and Sport
Locations (1):
- Friedrich-Alexander University Erlangen-Nürnberg, Department of Sport Science and Sport, Gebbertstr. 123b, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: project website — http://www.sport.fau.de/lehrstuehle-und-fachgebiete/bewegung-und-gesundheit/forschungsprojekte/optimierung-motorischer-lernprozesse-in-der-rehabilitation-von-parkinsonpatienten/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-19): https://cdn.clinicaltrials.gov/large-docs/90/NCT03886090/Prot_SAP_000.pdf